CLINICAL TRIAL: NCT03650270
Title: Childhood Convulsive Status Epilepticus - In Search Of Optimal Drug Management In A Resource Limited Setting
Brief Title: Childhood Convulsive Status Epilepticus Management In A Resource Limited Setting
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Cape Town (Other)
Responsible Party: Principal Investigator, Jo M Wilmshurst, Head of Department of Paediatric Neurology, Red Cross War Memorial Childrens Hospital, University of Cape Town
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 297/2005
Record Dates: First submitted 2018-08-17; First posted 2018-08-28 (Actual); Last update posted 2018-08-28 (Actual); Status verified 2018-08

CONDITIONS: Pediatric Status Epilepticus
MeSH Terms: interventions — Phenobarbital; Phenytoin; Midazolam

STUDY DESIGN:
Intervention Model Description: random allocation to 2 study protocols
Who Masked: Outcomes Assessor
Masking Description: The specific treatment protocol was blinded to the data analyser
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Phenobarbital (Experimental): If allocated to this arm 'Phenobarbital' (PHB group), the clinician gives an IV bolus of phenobarbital (20mg/kg ). If CSE did not terminate after 5 - 10 minutes, a second dose is given at half the dosage (10mg/kg) and a third dose (10mg/kg) is given if CSE persists 5-10 minutes after that.
  Interventions: Drug: Phenobarbital
- Phenytoin / Midazolam infusion (Active Comparator): In the 'Phenytoin / Midazolam infusion' (PHY/MDZ group), children are given a dose (20mg/kg) of IV phenytoin mixed with 50mL of normal saline solution and administered over 30 minutes . If the child is still in CSE 5-10 minutes after the phenytoin is given, they then start on a midazolam infusion. This includes a loading dose of IV midazolam (0.2mg/kg) followed by an infusion set at 3mg/kg into 50mL 5% dextrose water given at a rate of 1-4 mL/hour (equivalent to 1-4 mcg/kg/min ).
  Interventions: Drug: Phenobarbital

INTERVENTIONS:
Drug: Phenobarbital — Three repeated doses of pareneteral phenobarbital was compared to a single parenteral infusion of phenytoin followed by an infusion of parenteral midazolam
  Other Names: Phenytoin; Midazolam

SUMMARY:
Convulsive status epilepticus (CSE) is a potentially devastating condition which can result in significant morbidity and mortality. Studies addressing status epilepticus in children are rare and there is a paucity of large randomised controlled trials in children looking at forms of drug treatment for SE. There is consistency worldwide in guidelines for first line treatment of CSE with benzodiazepines, with slight variations in type and route of administration of agents. Second line therapy usually entails phenobarbital or phenytoin parenterally. Both repeated phenobarbital loading doses and midazolam infusions have been shown to be effective and safe in the management of established convulsive SE, but there are no prospective randomized controlled trials comparing the two in children.

Our study has been undertaken to review 2 existing, and routinely used, interventions for children presenting to our center with acute convulsive seizures. In order to permit comparable data to be collected we are randomly allocating these standard interventions prospectively. This is in order to compare the efficacy and safety of two treatment protocols (phenobarbital vs phenytoin and midazolam) both of which as stated are already part of existing standard protocols internationally and in South Africa. Parenteral phenobarbital is a safe, affordable and easy to use drug in the management of status epilepticus especially for poorly resourced communities where undertaking infusions may be unsafe, time consuming or unavailable.

We hypothesize that repeated phenobarbital loading is as effective and safe, or more so, than phenytoin followed by midazolam infusion in the management of established and refractory childhood convulsive SE. If proven, then the former would be a viable option for all health care workers with access to intravenous routes (including Day hospitals) where infusions are unsafe, time consuming or unavailable.

DETAILED DESCRIPTION:
This prospective study was conducted at the Red Cross War Memorial Children's Hospital (RCWMCH) and recruitment ran from between March 2015 to March 2018. All patients presenting with convulsive status epilepticus (CSE) who presented to the medical emergency unit at RCWMCH and needed therapeutic intervention were entered into the study by the attending medical staff. Study data was collected using REDCap hosted by the University of Cape Town's eResearch Centre and the study was approved by the UCT Human Research Ethics Council (UCT HREC 297/2005).

Definitions The definition of CSE was defined as any convulsive seizure that lasted longer than five minutes or multiple discrete seizures between which there is no extended period of recovery between events (Trinka et al., 2015). The onset of CSE was defined as the time provided by the caregiver who accompanied the child. The time to admission and to treatment were recorded by the staff in the unit. If children were admitted multiple times, each admission was captured independently, but only data from the first admission was included in this report . The full diagnosis of CSE was described using the multiaxial classification system. However, as it was not possible to perform EEG on all patients, this axes was excluded. Febrile status epilepticus was defined .

Treatment protocols Upon entry into the study, children were randomly allocated to one of two protocols . Both these protocols are well-established treatment protocols used in the sub-Saharan African setting for the management of SE . Randomization of protocols was performed using a free online platform (Research Randomizer ©). Both protocols began with children receiving first-line benzodiazepines (either midazolam, lorazepam or diazepam) which were either administered intravenously (IV), per rectally, intranasally or sublingually. If the children did not respond to single dose of benzodiazepines, they were given a second dose 5-10 minutes after the first dose. Pre-hospital administration of benzodiazepines by emergency services were counted if administered intravenously. However, all other routes of administration were not counted due to the lack of consistency in their administration.

If CSE continued after two doses of benzodiazepines, children were then randomized to second-line agents according to the protocol allocated to them. The one protocol, termed 'Phenobarbital' (PHB), instructed the clinician to give giving an IV bolus of phenobarbital (20mg/kg ). If CSE did not terminate after 5 - 10 minutes, a second dose was given at half the dosage (10mg/kg) and a third dose (10mg/kg) was given if CSE persisted 5-10 minutes after that.

In the second protocol, termed 'Phenytoin / Midazolam infusion' (PHY/MDZ), children were given a dose (20mg/kg) of IV phenytoin mixed with 50mL of normal saline solution and administered over 30 minutes . If the patient was still in CSE 5-10 minutes after the phenytoin was given, they were then started on a midazolam infusion. This included a loading dose of IV midazolam (0.2mg/kg) followed by an infusion set at 3mg/kg into 50mL 5% dextrose water given at a rate of 1-4 mL/hour (equivalent to 1-4 mcg/kg/min ).

If a patient child did not respond to the PHB or the PHY/MDZ protocols, they were referred to the pediatric intensive care unit (PICU). Other reasons for admission to the PICU included respiratory depression following administration of the second-line agent, need for inotropic support, etiology-related concerns requiring intensive monitoring (e.g. severe electrolyte imbalances) and or prolonged state of a depressed level of consciousness.

Demographic data inclusive of age, sex, etiologies, pre-existing medications, previous medical conditions and co-morbidities were recorded.

Outcome measures In comparing the two treatment protocols, we will only focused on the short-term outcomes of the children in each treatment protocol. These include how the agents affected the children's physiology, admission to PICU, whether subsequent breakthrough seizures occurred and days admitted to hospital. In measuring the effects on the children's physiology, their we will calculate heart rate, respiratory rate and mean arterial pressure from during CSE to immediately post-ictal period. This will be done by subtracting the first measurement as the child presented to the unit from the first measurement taken immediately after the child had stopped convulsing.

Data analysis During the analysis, the investigator performing the analysis was blinded to which protocol the patients children were allocated to. Group allocations will only be unblinded after statistical analysis is completed and verified by an external party. Data will analysed using SPSS Statistics (IBM Corp. Released 2016, Version 24.0. Armonk, NY: IBM Corp). Statistical measurements will be performed using both SPSS Statistics and GraphPad Prism version 6.0 (GraphPad Software, USA). For continuous data normality will be established using the Shapiro-Wilk test and thereafter parametric (i.e. paired or unpaired student's t-tests) or nonparametric tests (i.e. Mann-Whitney U test or Wilcoxon signed-rank test) will be performed. Normally distributed data will be reported as mean standard deviation. Data that is not normally distributed will be reported as median with the interquartile range (IQR). Categorical data will be summarized in contingency tables with differences between groups being identified using the Fisher-exact or chi-squared (X2) tests and associations calculated using odds ratios (OR). Significance will be defined as a p < 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Children in convulsive status epilepticus (as defined by Trinka et al 2015)

Exclusion Criteria:

* Children not in convulsive status epilepticus

Ages: 1 Month to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 198 (Actual)
Dates: Start 2015-03-01 (Actual); Primary Completion 2018-03-01 (Actual); Study Completion 2018-03-01 (Actual)

PRIMARY OUTCOMES:
Differences in anticonvulsant efficacy between different second-line anticonvulsant treatment protocols | Up to 24 hours from the time the patient was admitted.
  Assessing the time taken to reach seizure arrest after second-line agents given

SECONDARY OUTCOMES:
Differences in how patients tolerate each of the two second-line anticonvulsant treatment protocols | Up to 24 hours from the time the patient was admitted.
  Assessing differences physiological response to second-line anticonvulsant protocols
Differences in need for pediatric intensive care between the two second-line anticonvulsant protocols | Up to 24 hours from the time the patient was admitted.
  Assessing differences in proportion of patients who received second-line anticonvulsant therapy and then require admission to the pediatric intensive care unit
Differences in admission time between patients who receive on of the two second-line anticonvulsant protocols | For the full duration the patient is admitted, which on average is up to one full week (seven days).
  Assessing differences in the number of days the patient is admitted following admission

CONTACTS AND LOCATIONS:
Locations (1):
- Red Cross War Memorial Children's Hospital, Cape Town, Western Cape, South Africa

IPD SHARING:
Plan to Share IPD: Undecided
We are exploring what data would of use

REFERENCES:
- [Derived] Burman RJ, Ackermann S, Shapson-Coe A, Ndondo A, Buys H, Wilmshurst JM. A Comparison of Parenteral Phenobarbital vs. Parenteral Phenytoin as Second-Line Management for Pediatric Convulsive Status Epilepticus in a Resource-Limited Setting. Front Neurol. 2019 May 15;10:506. doi: 10.3389/fneur.2019.00506. eCollection 2019. PMID 31156538